CLINICAL TRIAL: NCT03369509
Title: Etude de Cohorte Des Patients Suivis en Allergologie au CHU de Grenoble : hypersensibilité Allergique et hypersensibilité Non Allergique
Brief Title: Allergic Versus Non Allergic Hypersensitivity Drug Reaction (BdDAllergo)
Acronym: BdDAllergo
Status: Terminated | Type: Observational
Why Stopped: departure of the investigator from the CHU Grenoble Alpes
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.038; 2017-A00378-45 (Other: ID RCB)
Record Dates: First submitted 2017-08-18; First posted 2017-12-12 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Allergic Hypersensitivity Drug Reaction Versus Non-allergic Hypersensitivity Drug Reaction Cross Reaction
Keywords: Drug hypersensitivity, drug allergy, cross reaction
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hypersensitivity drug reaction: Patient followed in the allergology department for the realization of immunoallergological test after suspicion of hypersensitivity drug reaction.

SUMMARY:
The creation of a database containing the medical data of patients followed in allergology at the University Hospital of Grenoble will permit to study allergic versus non-allergic hypersensitivity drug reaction as well as the risk of cross-reactions between medicinal drugs belonging to the same pharmacological class.

The main objectives of the study are to estimate and to compare the proportion of allergic hypersensitivity drug reaction and the proportion of non allergic hypersensitivity drug reaction, and to characterize these two types of hypersensitivity drug reaction on clinical, biological and chronological aspects.

In a second time, ancillary study will be conducted in order to :

* identify drugs that potentially induced histamine-liberation in patients diagnosed with non allergic hypersensitivity drug reaction
* investigate the risk of cross-reactions between drugs belonging to the same pharmacotherapeutic class in patients diagnosed with allergic hypersensitivity drug reaction.

DETAILED DESCRIPTION:
This study is an observational cohort study conducted at University Hospital of Grenoble. It include retrospectively and prospectively the patients followed in the allergology department for the realization of immunoallergological test after suspicion of hypersensitivity drug reaction. The data are collected in a database from medical consultation reports that are systematically reported to the pharmacovigilance regional center. An anonymization number is assigned for each patient included in the study.The data collected include patient's personal and family medical history, a clinical, biological and chronological description of the hypersensitivity reaction, the results of the immunoallergologic skin tests as well as the final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Cases where a non-iatrogenic cause was finally identified

Exclusion Criteria:

* For the estimation and comparison of the proportions, the patients who haven't carried out all their immunoallergologic tests investigations at the University Hospital of Grenoble are not included (this concerns patient who have realized only oral rechallenge test at hospital)
* To realize the comparative analysis of allergic versus non-allergic hypersensitivity drug reaction : cases that are insufficiently documented on clinical, biological and / or chronological aspects are excluded. This concerns especially patients who realize immunoallergologic tests investigations after a skin reaction that occurred "in childhood".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who realize a complete immunoallergologic tests investigations at the University Hospital of Grenoble.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Allergic Versus Non Allergic Hypersensitivity Drug Reaction | Through study completion, an average of 5 years
  Conclusion of the immunoallergologic tests investigations :
  * allergic hypersensitivity drug reaction case are diagnosed when the skin tests are positive or the skin tests are negative but the oral rechallenge test is positive.
  * non allergic hypersensitivity drug reaction case are diagnosed when the skin tests are negative AND the oral rechallenge test is negative.

SECONDARY OUTCOMES:
- To determine the proportion of drugs involved in in allergic hypersensitivity drug reaction for each pharmacotherapeutic class | Through study completion, an average of 5 years
  Immunoallergologic tests investigations that conclude to an allergic hypersensitivity drug reaction
immediate allergic hypersensitivity and delayed allergic hypersensitivity on clinical, biological and chronological aspects | Through study completion, an average of 5 years
  Conclusion of the immunoallergologic tests investigations :
  * immediate allergic hypersensitivity drug reaction case are diagnosed when the skin tests are positive at 20 minutes for Prick tests or IDR or the skin tests are negative but the oral rechallenge test is positive immediately.
  * delayed allergic hypersensitivity drug reaction case are diagnosed when the skin tests are positive at 24 or 48 hours for IDR or the skin tests are negative but the oral rechallenge test is positive in the days following the reintroduction of treatment.
To determine the proportion of drugs that potentially induced histamine-liberation in patients diagnosed with non allergic hypersensitivity drug reaction for each pharmacotherapeutic class | Through study completion, an average of 5 years
  Conclusion of the immunoallergologic tests investigations :
  - non allergic hypersensitivity drug reaction case are diagnosed when the skin tests are negative AND the oral rechallenge test is negative.
- Proportion of cross-reaction between drugs belonging to the same pharmacotherapeutic class in patients diagnosed with allergic hypersensitivity drug reaction. | ancillary study, Through study completion, an average of 5 years
  Conclusion of the immunoallergologic tests investigations :
  - Cross-reaction are diagnosed when the immunoallergologic test investigation is positive for medicinal products belonging to the same pharmacotherapeutic class as the responsible treatment of the skin reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nassima YAHIAOUI, Principal Investigator — UniversityHospital Grenoble
Locations (1):
- UniversityHospitalGrenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cousin F, Catelain A, Philips K, Favier B, Queuille E, Nicolas JF. [Immediate hypersensitivity is rarely implicated in drug induced urticaria]. Ann Dermatol Venereol. 2003 Mar;130(3):321-4. French. PMID 12746667
- [Result] Ponvert C, Scheinmann P. [Allergic and pseudo-allergic reactions to betalactam antibiotics]. Arch Pediatr. 2003 Jul;10(7):658-65. doi: 10.1016/s0929-693x(03)00272-0. No abstract available. French. PMID 12907084
- [Result] Nosbaum A, Pralong P, Rozieres A, Dargaud Y, Nicolas JF, Berard F. [Delayed-type hypersensitivity to heparin: diagnosis and therapeutic management]. Ann Dermatol Venereol. 2012 May;139(5):363-8. doi: 10.1016/j.annder.2012.01.017. Epub 2012 Mar 9. French. PMID 22578340